CLINICAL TRIAL: NCT01580566
Title: Renal Structural, Functional and Cytokine Responses to Acute Myocardial Injury in Man
Brief Title: Renal Acute MI Study
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Seniour Lecturer, Monash University
Other Study IDs: CP-03/11
Record Dates: First submitted 2012-04-12; First posted 2012-04-19 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Infarction; Kidney Function
Keywords: Myocardial Infarction (MI); Kidney function; bio-markers
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to measure bio-markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1 - Control: Non-Q wave MI subjects with normal cardiac and renal function (defined as eGFR >60ml/min) not undergoing a cardiac procedure involving contrast will serve as "control" for renal injury subjects.
- Group 2 - stable CAD or non-Q wave MI: Patients undergoing coronary angiography +/- PCI for stable CAD or non-Q wave MI with normal cardiac and renal function (defined as eGFR >60ml/min) will control for the contrast STEMI patients are likely to receive as part of their post-MI management
- Group 3 - Acute STEMI without chronic kidney disease: Acute STEMI patients (n=40), without chronic kidney disease (defined as eGFR ≥60ml/min).
- Group 4 - Acute STEMI with kidney disease: Acute STEMI patients (n=40), with evidence of background chronic kidney disease (eGFR <60ml/min).

SUMMARY:
The purpose of this study is to determine if a sizable myocardial infarction (heart attack) results in negative changes to renal structure and function (i.e. has a negative impact on the kidneys).

To determine if the renal response to a myocardial infarction is a predictor of the patients future health.

DETAILED DESCRIPTION:
Chronic heart and kidney disease are increasingly common in Western society. Both conditions are associated with frequent hospitalisation and increased mortality. Furthermore, there are mechanistic reasons why one condition may beget the other; the so-called "cardiorenal syndrome". The investigators therefore wish to determine if a sizable myocardial infarction (heart attack) results in negative changes to renal structure and function (i.e. has a negative impact on the kidneys). The investigators also wish to determine if the renal response to a myocardial infarction is a predictor of the patients future health. To do this the investigators will measure markers of kidney function at the time of the heart attach, at discharge, 1 month, 6 months and 12 months and correlate this with the patients clinical condition.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years

Have provided written informed consent

Group 1:

* Non-Q wave MI patients
* normal cardiac and renal function
* No use of contrast
* eGFR > 60ml/min

Group 2:

* Patients undergoing coronary angiography +/- PCI for stable CAD or non-Q wave MI
* normal cardiac and renal function
* eGFR > 60ml/min

Group 3:

* Acute STEMI Full thickness infarct (STEMI)
* eGFR ≥ 60ml/min

Group 4:

* Acute STEMI Full thickness infarct (STEMI)
* eGFR < 60ml/min

Exclusion Criteria:

* Unable or unwilling to comply with the study protocol
* Underlying medical condition which, in the opinion of the investigator, will effect the safely or efficacy of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have presented to the Emergency Department with chest pain caused by a possible myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
changes in renal function and structure | Baseline, discharge, 1 month, 6 months and 12 months

SECONDARY OUTCOMES:
renal response to myocardial infarction | baseline, discharge, 1 month, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Alfred Hospital/Monash.University; Henry Krum, MBBS FRACP PhD, Principal Investigator — Alfred Hospital/Monash University
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia